CLINICAL TRIAL: NCT07377227
Title: Evaluation of Social Cognition: A New Screening Approach for Autism
Brief Title: Social COgnition Screening
Acronym: ECoS-A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2025_843_0181
Record Dates: First submitted 2025-11-17; First posted 2026-01-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Eye-tracking; Autism Spectrum Disorder; Social Cognition; Diagnosis
Keywords: Eye-tracking; Autism Spectrum Disorder; Social Cognition; Diagnosis
MeSH Terms: conditions — Autism Spectrum Disorder; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Spectrum Disorder (Experimental): Autism Spectrum Disorder
  Interventions: Other: eye-tracking; Other: cognitive assessments
- typically developing peers (Active Comparator): typically developing (TD) peers
  Interventions: Other: eye-tracking; Other: cognitive assessments

INTERVENTIONS:
Other: eye-tracking — eye-tracking
Other: cognitive assessments — cognitive assessments

SUMMARY:
Social cognition refers to the mental processes involved in social interactions, including social perception, motivation, communication, emotion recognition, and theory of mind. Face perception plays a key role in children's social development, but children with Autism Spectrum Disorder (ASD) tend to look less at social stimuli, especially faces, than typically developing (TD) peers. Eye-tracking studies highlight these visual exploration differences, linked to difficulties in joint attention, emotion recognition, and theory of mind, as well as in executive and memory functions. Standard diagnostic tests often require active participation and sufficient language, which makes assessment challenging for children with ASD and additional cognitive or language impairments.

This research project investigates how visual activity supports social cognition depending on cognitive and language levels, hypothesizing that eye-tracking can provide useful indicators for ASD screening and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* ASD Group:
* Boys or girls diagnosed with Autism Spectrum Disorder (based on clinical tools and observations)
* Aged between 4 and 10 years old
* Affiliation with a social security scheme
* Informed consent of those with parental authority
* DT Group:
* Boys or girls
* Aged between 4 and 10
* Attending school in the Hauts-de-France region
* Affiliation with a social security scheme
* Consent of those with parental authority

Exclusion Criteria:

* For ASD: Uncorrected visual or auditory impairments.
* For DT: Intellectual disability, neurological or genetic disorders, autistic traits reported by teachers. The discrepancy between actual age and abilities calculated on the basis of standardised test scores

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
differences in visual exploration patterns between both groups | 2 years
  Differences in visual exploration patterns between both groups Visual exploration patterns are determined with TOM Test Battery, PPVT-5, Raven's 2 and FEE tests
Classification performance of machine learning algorithms in distinguishing ASD from TD | 2 years
  Classification performance of machine learning algorithms in distinguishing ASD from TD

SECONDARY OUTCOMES:
Correlations between eye-tracking measures and cognitive scores | 2 years
  Eye-tracking patterns are determined with TOM Test Battery, PPVT-5, Raven's 2 and FEE tests
Developmental trajectory analysis in TD children | 2 years
Identification of cognitive subgroups within ASD group | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No